CLINICAL TRIAL: NCT04320368
Title: China National Clinical Research Center Alzheimer's Disease and Neurodegenerative Disorder Research
Brief Title: China Alzheimer's and Neurodegenerative Disorder Research
Acronym: CANDOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Shiping Li, Principle Investigator, Beijing Tiantan Hospital
Other Study IDs: Z181100001518005
Record Dates: First submitted 2020-03-10; First posted 2020-03-25 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Impairment
Keywords: Alzheimer's disease; vascular cognitive impairment; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, urine and feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alzheimer's disease cohort: 1. Aged 40-100 years old (≥ 40 years old, ≤ 100 years old).
  2. Diagnosed with AD according to Alzheimer disease diagnostic criteria following NINCDS-ADRDA 1984 or NIA-AA 2011 guideline.
  3. Had adequate hearing, vision and comprehension and verbal expression to complete the cognitive assessments.
  4. Had at least 3 years of education.
  5. Signed informed consent.
- Post-stroke cognitive observation cohort: 1. Aged 40-100-years old (≥ 40 years old, ≤ 100 years old).
  2. Cerebral infarction is diagnosed according to World Health Organization diagnostic criteria and was the first symptomatic onset.
  3. The time from onset to enrollment was less than 7 days.
  4. Had adequate hearing, vision and comprehension and verbal expression to complete the cognitive assessments.
  5. Had at least 3 years of education.
  6. Signed informed consent.
- A cohort of people with normal cognitive function: 1. Aged 40-100 years old (≥ 40 years old, ≤ 100 years old).
  2. The patients are cognitively normal and able to live and work independently
  3. Had adequate hearing, vision and comprehension and verbal expression to complete the cognitive assessments.
  4. Had at least 3 years of education.
  5. Signed informed consent.

SUMMARY:
This is a multi-center study that has three cohorts: 1) cognitive normal cohort (CN), 2) Alzheimer's disease cohort (AD) and 3) vascular cognitive impairment cohort (VCI). The goal of this study is to understand the risk factors of AD and VCI and to identify high risk patients for early intervention. It will collect demographic information, family history, medical history, neuropsychological tests, imaging studies and biological samples through standard and uniform procedures.

DETAILED DESCRIPTION:
In this prospective study, we will recruit subjects into one of the three groups based on inclusion and exclusion criteria: 1) CN, 2) AD and 3) VCI. We will follow up with each of them subject at designated time points up to 2 years. We will collect demographic, medical, imaging (MRI and PET scans), genetic information and various biological samples (blood, saliva, urine and feces) during the study period. This study uses a case-control study design. The matched cases will have similar age, gender and education levels. By studying the relationship between risk factors of AD and VCI, we will establish norms and parameters in the Chinese population.

ELIGIBILITY:
1. The inclusion and exclusion criteria of AD group.

   1.1 The AD group inclusion criteria: 1.1.1 Aged 40-100 years old (≥ 40 years old, ≤ 100 years old). 1.1.2 Diagnosed with AD according to Alzheimer disease diagnostic criteria following NINCDS-ADRDA1984 or NIA-AA 2011 guideline.

   1.1.3 Had adequate hearing, vision and comprehension and verbal expression to complete the cognitive assessments.

   1.1.4 Had at least 3 years of education. 1.1.5 Signed informed consent.

   1.2 The AD group exclusion criteria: 1.2.1 Sequelae after previous history of severe central nervous system infection, multiple sclerosis, autoimmune encephalitis, Hashimoto's encephalopathy, etc.

   1.2.2 Previous history of instable epilepsy. 1.2.3 Systemic diseases affect the central nervous system (CNS), such as abnormal liver and kidney functions.

   1.2.4 History of hereditary diseases that affect cognitive function (such as Huntington's disease, Down's syndrome, CADASIL, adrenal leukodystrophy, mitochondrial encephalopathy, etc.).

   1.2.5 Infection and immune-related diseases affecting the central nervous system (systemic lupus erythematosus, undertreated HIV infection or a history of CNS syphilis infection, etc.).

   1.2.6 Metabolic and endocrine disorders (requiring new treatment or adjustment of current treatment for thyroid dysfunction, folate or vitamin B12 deficiency).

   1.2.7 Had contraindications for MRI (e.g., pacemakers, stents, claustrophobia.) or did not cooperate with PET scans.
2. The inclusion and exclusion criteria of post-stroke cognitive observation group.

   2.1 The inclusion criteria of post-stroke cognitive observation group: 2.1.1 Aged 40-100-years old (≥ 40 years old, ≤ 100 years old). 2.1.2 Cerebral infarction is diagnosed according to World Health Organization diagnostic criteria13 and was the first symptomatic onset.

   2.1.3 The time from onset to enrollment was less than 7 days. 2.1.4 Had adequate hearing, vision and comprehension and verbal expression to complete the cognitive assessments.

   2.1.5 Had at least 3 years of education. 2.1.6 Signed informed consent.

   2.2 The exclusion criteria of post-stroke cognitive observation group: 2.2.1 Prior to the onset of acute infarction had no conditions known to affect cognitive function, such as vascular dementia, dementia with Lewy body dementia, frontotemporal dementia, Parkinson's disease dementia, epilepsy, stroke, hydrocephalus, multiple sclerosis, traumatic brain injuries, genetic disorders affecting cognition, alcoholism, uncontrolled depression or other psychiatric disorders and Alzheimer's disease and IQCODE>3.5.

   2.2.2 Sequelae after previous history of severe central nervous system infection, multiple sclerosis, autoimmune encephalitis, Hashimoto's encephalopathy, etc.

   2.2.3 Previous history of instable epilepsy. 2.2.4 Systemic diseases affect the CNS, for abnormal liver and kidney functions.

   2.2.5 History of hereditary diseases that affect cognitive function (such as Huntington's disease, down syndrome, CADASIL, adrenal leukodystrophy, mitochondrial encephalopathy, etc.).

   2.2.6 Infection and immune-related diseases affecting the central nervous system (systemic lupus erythematosus, undertreated HIV infection or a history of CNS syphilis infection, etc.).

   2.2.7 Metabolic and endocrine disorders (requiring new treatment or adjustment of current treatment for thyroid dysfunction, folate or vitamin B12 deficiency).

   2.2.8 Reject or had contraindications for MRI (e.g., pacemakers, stents, claustrophobia.).
3. The inclusion and exclusion criteria of normal cognitive group.

3.1 The inclusion criteria of normal cognitive group: 3.1.1 Aged 40-100 years old (≥ 40 years old, ≤ 100 years old). 3.1.2 The patients are cognitively normal and able to live and work independently.

3.1.3 Had adequate hearing, vision and comprehension and verbal expression to complete the cognitive assessments.

3.1.4 Had at least 3 years of education. 3.1.5 Signed informed consent.

3.2 The exclusion criteria of normal cognitive group: 3.2.1 The patients had no conditions known to affect cognitive function, such as vascular dementia, dementia with Lewy body dementia, frontotemporal dementia, Parkinson's disease, epilepsy, stroke, hydrocephalus, multiple sclerosis, traumatic brain injuries, genetic disorders affecting cognition, alcoholism, uncontrolled depression or other psychiatric disorders, Parkinson's disease, epilepsy or Alzheimer's disease.

3.2.2 Sequelae after previous history of severe central nervous system infection, multiple sclerosis, autoimmune encephalitis, Hashimoto's encephalopathy, etc.

3.2.3 Previous history of instable epilepsy. 3.2.4 Systemic diseases affect the CNS, for abnormal liver and kidney functions.

3.2.5 History of hereditary diseases that affect cognitive function (such as Huntington's disease, down syndrome, CADASIL, adrenal leukodystrophy, mitochondrial encephalopathy, etc.).

3.2.6 Infection and immune-related diseases affecting the central nervous system (systemic lupus erythematosus, undertreated HIV infection or a history of CNS syphilis infection, etc.).

3.2.7 Metabolic and endocrine disorders (requiring new treatment or adjustment of current treatment for thyroid dysfunction, folate or vitamin B12 deficiency).

3.2.8 Reject or had contraindications for MRI (e.g., pacemakers, stents, claustrophobia.).

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alzheimer's disease cohort and post-stroke cognitive observation cohort will be recruited from participating hospitals.
  Cognitively normal cohort will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Data records | 4-5 years
  We will record the number of participants at several follow-up visits, the basic condition at the follow-up. If the visit is not completed, record the cause of this loss.
  At baseline, record the demographic information, past medical history and medication history, vital signs and neuropsychological scales. The PET-CT scan were recorded during the 4-year visit. Collect the results of cerebral MRI, laboratory tests and neuropsychological scales of all participants at baseline, 12, 24, 36 and 48 months and biological samples. For VCI cohort, we will record the basic conditions and partial neuropsychological scales at 3-month and 6-month follow-up.
Neuropsychological scales | 4-5 years
  Mini-Mental State Examination (MMSE), Montreal-Cognitive Assessment (MoCA), the Geriatric Depression Scale (GDS), The Activities of Daily Living Questionnaire(ADL), Digit Span Memory Test, Rey Auditory Verbal Learning Test (RAVLT), Rey-Osterrieth Complex Figure Test(ROCF), Trail Making Test A and B, Stroop test, Verbal Fluency Test, Boston Naming Test, Clock-Drawing Test, Narcissism Test (NPI), Symbol Digit Modalities Test(SDMT), Clinical Dementia Rating (CDR)

CONTACTS AND LOCATIONS:
Overall Officials: Shiping Li, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All data are available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available at one year after the study completion.
Access Criteria: Committee review

REFERENCES:
- [Background] Prince MJ, Wu F, Guo Y, Gutierrez Robledo LM, O'Donnell M, Sullivan R, Yusuf S. The burden of disease in older people and implications for health policy and practice. Lancet. 2015 Feb 7;385(9967):549-62. doi: 10.1016/S0140-6736(14)61347-7. Epub 2014 Nov 6. PMID 25468153
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Derived] Wang Y, Wang Q, Tong L, Zheng H, Wang Y, Li S. U-shaped association between post-stroke cognitive impairment and high-density lipoprotein cholesterol at the acute period of stroke. Arch Gerontol Geriatr. 2025 Dec;139:106002. doi: 10.1016/j.archger.2025.106002. Epub 2025 Aug 26. PMID 40915091
- [Derived] Wang Q, Wang Y, Li S, Shi J. PACAP-Sirtuin3 alleviates cognitive impairment through autophagy in Alzheimer's disease. Alzheimers Res Ther. 2023 Oct 27;15(1):184. doi: 10.1186/s13195-023-01334-2. PMID 37891608
- [Derived] Wang Y, Wang S, Zhu W, Liang N, Zhang C, Pei Y, Wang Q, Li S, Shi J. Reading activities compensate for low education-related cognitive deficits. Alzheimers Res Ther. 2022 Oct 14;14(1):156. doi: 10.1186/s13195-022-01098-1. PMID 36242017